CLINICAL TRIAL: NCT03378310
Title: A Randomized, Open-Label Study to Evaluate the Bioavailability of a BMS-986205 Tablet Containing Free Base Relative to a Reference Tablet in Healthy Participants
Brief Title: A Study in Healthy Participants Evaluating the Absorption of a BMS-986205 Tablet Into the Bloodstream Compared to a Reference Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CA017-069
Record Dates: First submitted 2017-12-15; First posted 2017-12-19 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — linrodostat

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Reference tablet followed by BMS-986205 tablet with free base (Experimental): BMS-986205 reference tablet (treatment period 1) followed by BMS-986205 tablet with free base (treatment period 2).
  Interventions: Drug: BMS-986205 reference tablet; Drug: BMS-986205 tablet with free base
- BMS-986205 tablet with free base followed by reference tablet (Experimental): BMS-986205 tablet with free base (treatment period 1) followed by BMS-986205 reference tablet (treatment period 2).
  Interventions: Drug: BMS-986205 reference tablet; Drug: BMS-986205 tablet with free base

INTERVENTIONS:
Drug: BMS-986205 reference tablet — Single, 100 mg oral dose.
Drug: BMS-986205 tablet with free base — Single, 100 mg oral dose.

SUMMARY:
This is a Phase 1, open-label, randomized study in healthy participants to evaluate the absorption of a BMS-986205 tablet into the bloodstream compared to a reference tablet. Eligible participants will be randomly assigned to 1 of 2 treatment sequences and will receive a single, oral dose of BMS-986205 twice over 22 days. Participants must remain at the clinical facility for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Signed, written informed consent.
* Healthy male and female participants (not of childbearing potential), determined by medical history, physical examination, electrocardiograms (ECGs) and clinical laboratory tests.
* Normal renal (kidney) function.
* Body Mass Index (BMI) of 18.0 kg/m2 to 32.0 kg/m2, inclusive.
* Women must have documented proof they are not of childbearing potential.
* Males who are sexually active with women of childbearing potential must agree to follow instructions for method(s) of contraception for the duration of treatment and 110 days after the last dose of BMS-986205. In addition, male participants must be willing to refrain from sperm donation during this time.

Exclusion Criteria:

* Women of childbearing potential or breastfeeding.
* Active tuberculosis (TB) requiring treatment or documented latent TB within the previous 3 years. Also excluded are participants with evidence of a past TB infection without documented adequate therapy.
* History of pulmonary, renal, or liver disease; or of cardiac arrhythmias.
* Recent (within 6 months of study drug administration) history of smoking or current smokers. This includes participants using electronic cigarettes or nicotine-containing products such as tobacco for chewing, nicotine patches, nicotine lozenges or nicotine gum.
* Donation of blood to a blood bank or in a clinical study (except screening or follow-up visit) within 4 weeks of study drug administration (within 2 weeks for plasma only).

Other protocol defined inclusion/exclusion criteria could apply.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-02-22 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of BMS-986205 tablet with free base compared to reference tablet. | Up to Day 22
  Measured by plasma concentration.
Area under the plasma concentration time curve from time zero to 168 hours after dosing (AUC[0-168]) of BMS-986205 tablet with free base compared to reference tablet. | Up to Day 22
  Measured by plasma concentration.

SECONDARY OUTCOMES:
Incidence of non-serious Adverse Events (AEs). | Up to Day 22
  Safety and tolerability as measured by incidence of non-serious AEs.
Incidence of Serious Adverse Events (SAEs). | Up to Day 22
  Safety and tolerability as measured by incidence of SAEs.
Incidence of Adverse Events (AEs) leading to discontinuation. | Up to Day 22
  Safety and tolerability as measured by incidence of AEs leading to discontinuation.
Number of participants with vital sign abnormalities. | Up to Day 22
Number of participants with electrocardiogram (ECG) abnormalities. | Up to Day 22
Number of participants with clinical laboratory abnormalities. | Up to Day 22
Number of participants with physical examination abnormalities. | Up to Day 22

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- PPD Austin Clinic, Austin, Texas, United States

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/Recalls/
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/pages/investigator_inquiry_form.aspx